CLINICAL TRIAL: NCT05998551
Title: Effectiveness of Single Shot Intra-thecal Analgesia in Multiparous Women Scheduled for Normal Vaginal Delivery.
Brief Title: Single Shot Intrathecal Analgesia in Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: intra-thecal analgesia
Record Dates: First submitted 2023-06-16; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-05

CONDITIONS: Effectiveness of Single Shot Intra-thecal Analgesia in Multiparous Women Scheduled for Normal Vaginal Delivery
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Bupivacaine

STUDY DESIGN:
Intervention Model Description: The eligible parturients will be randomly allocated into three groups according to the additive added to a fixed dose of local anesthetic (1ml=5mg of 0.5% hyperbaric bupivacaine).Total volume of 2 ml will be given to each patient
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computer generated number lists and use of sealed opaque envelopes , double blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine Group (Active Comparator): participants will receive intrathecal injection of 5mg (1ml) of 0.5% hyperbaric bupivacaine + 1 ml contain 5μg dexmedetomidine(0.05ml dexmedetomidine in insulin syringe+ 0.95ml normal saline).
  Interventions: Drug: Dexmedetomidine
- Fentanyl group (Active Comparator): participants will receive intrathecal injection of 5 mg (1ml) of 0.5% hyperbaric bupivacaine + 1 ml contain 12.5μg fentanyl(0.25ml fentanyl in insulin syringe+ 0.75ml normal saline).
  Interventions: Drug: Fentanyl
- Control group (Active Comparator): participants will receive intrathecal injection of 5mg (1ml) of 0.5% hyperbaric bupivacaine + 1 ml normal saline
  Interventions: Drug: Bupivacaine Hcl 0.5% Inj

INTERVENTIONS:
Drug: Dexmedetomidine — intrathecal injection of dexmedetomidine added to hyperbaric bupivacaine
  Arms: Dexmedetomidine Group
Drug: Fentanyl — intrathecal injection of fentanyl added to hyperbaric bupivacaine
  Arms: Fentanyl group
Drug: Bupivacaine Hcl 0.5% Inj — intrathecal injection of hyperbaric bupivacaine only
  Arms: Control group

SUMMARY:
Effectiveness of single shot intra-thecal analgesia in multiparous women scheduled for normal vaginal delivery

DETAILED DESCRIPTION:
Labor is a physiological and natural process, as well as a complicated and subjective experience.Except for a few women, childbirth is unquestionably a painful experience. Women's understanding of delivery's pain is influenced by various factors, making each experience special. As opposed to other painful life events, labor pain consistently ranks high on the pain rating scale.

In this study ,the investigators are going to investigate the effectiveness and safety of intrathecal analgesia for labour using bupivacaine with fentanyl or dexmedetomidine.

ELIGIBILITY:
* Inclusion criteria:

  * Multiparous women who received antenatal care, presented for vaginal delivery of uncomplicated term pregnancy of singleton fetus with engaged fetal head and cervical dilatation of at least 5 cm requiring oxytocin augmentation, and requested analgesia.
  * Age: patients between 22-45 years old.
* Exclusion criteria:

  * Refusal of procedure or participation in the study.
  * Patients with pre-existing or pregnancy-induced hypertension, abnormal fetal heart rate tracings, obesity, endocrinal diseases and/or diagnosed fetal abnormalities.
  * Contraindication to neuraxial block.
  * Allergy to any of the study drugs.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Duration of pain relief | Up to 6 hours after intrathecal injection
  The duration of pain relief will be defined as the duration from intrathecal injection till the VAS became more than 4
analgesic onset time | within 15 minutes after intrathecal injection
  The analgesia onset time will be defined as the time from intrathecal injection until the VAS became less than 4
maximum level of sensory block | 15 min after the intrathecal injection
  Temperature will be assessed using methylated soaked swabs on both sides of the body
visual analogue scale (VAS) of the labour pain | 6 hours after intrathecal injection
  The VAS (ranging from 0 = pain-free up to 10 = worst imaginable pain) of the labour pain will be recorded before the intrathecal injection, every 5 min for the first 20 min, then every 30 min for 6 hours
S1 regression time | 6 hours after intrathecal injection
  S1 regression time will be defined as the time from intrathecal injection to sensory regression to S1 dermatome

SECONDARY OUTCOMES:
Maternal blood pressure | 6 hours post operative
  any change more than 20% of baseline mean arterial pressure
Maternal heart rate | 6 hours post operative
  any change more than 20% of baseline heart rate
Post operative nausea and vomiting | 6 hours post operative
  Number of participants having post operative nausea and vomiting
Post operative urinary retention | 6 hours post operative
  Number of participants having post operative urinary retention
Fetal heart sounds | from intrathecal injection till delivery
  Change more than 20% of fetal heart sounds before delivery
Fetal APGAR score | till 5 minutes after delivery
  APGAR score (1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2 at 1 and 5 minutes after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided